CLINICAL TRIAL: NCT06636253
Title: Does Stress Change EEG Measures in Students: A Feasibility Study.
Acronym: EEG_stress
Status: Recruiting | Type: Observational
Sponsor: Scotland College of Chiropractic (Other)
Responsible Party: Principal Investigator, Alice Cade, Senior lecturer and research fellow, Scotland College of Chiropractic
Other Study IDs: 348503
Record Dates: First submitted 2024-09-12; First posted 2024-10-10 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Electroencephalogram; Stress
Keywords: Electroencephalogram; stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SCC students: Healthy adults attending and actively enrolled in the Scotland College of Chiropractic's degree program and who were without health issues or mental disorders.

SUMMARY:
Psychological stress is a frequent human affection and has a considerable impact on modern society, and tertiary-level students often report increased stress levels as the semester progresses. While many questionnaires assess psychological stress, they do not capture objective data. Much research has shown that electroencephalography (EEG) can capture objective markers of stress, and recent studies have shown that EEG can even classify stress levels.

This study aims to assess the feasibility of using EEG to objectively assess stress over the course of a semester of work in chiropractic students engaged in a Masters level course in Scotland.

DETAILED DESCRIPTION:
The study's primary aim is to assess the feasibility of a more extensive future study. The investigators also hypothesise that as the semester progresses, participants will exhibit changes in their EEG outcomes that may be related to longitudinal or direct stressors.

Study design and setting This study will be an observational study with a stress-related questionnaire (Depression, Anxiety, and Stress Scale - 21 (DASS-21)) over three time-points.

Participants The investigators aim to recruit 10 participants and assess them three times over the course of their semester, early, middle, and late semester, with at least a four-week gap between each data collection. The investigators aim to recruit only healthy Scottish chiropractic students with no prior diagnosed mental disorder and who are capable of understanding the study procedure.

Procedure Following screening for eligibility and consent, i.e., visit one (baseline), participants will be asked to answer a questionnaire and undergo EEG measurement and Montreal imaging stress task (MIST). The same EEG and questionnaire procedure will be performed in the remaining two data collection sessions.

Each EEG recording session, with the participant seated, will consist of a two-minute resting state with the eyes closed for a baseline relaxation level among the participants. A following two-minute eyes-open phase will take place. After which, participants will be asked to perform the experimental phase of the MIST task, a following two-minute recording phase will be with the eyes open, and a final two-minute resting phase with eyes closed will conclude the task.

The investigators aim to conclude the data collection around 16 weeks after the initial participant is recruited.

ELIGIBILITY:
Inclusion Criteria:

Healthy Scottish chiropractic students with no prior diagnosed mental disorder and who are capable of understanding the study procedure.

Exclusion Criteria:

A pre-diagnosed mental health disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Scottish chiropractic college students
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility recruitment rates | 0, 6, 12 weeks
  recruitment rates - how many people were recruited ove rthe study time period
Feasibility - retention | 0, 6, 12 weeks
  Participant retention - how many participants completed the full study
Feasibility - queries | 12 weeks
  queries from participants - how many question did participants ask and were they answerable
Feasibility - ease | 12 weeks
  Ease of data collection - was the data collection procedure manageable for the investigator
Feasibility - Adverse | 12 weeks
  Adverse events - were any adverse events either minor or significant, recorded at any time throughout the trial

SECONDARY OUTCOMES:
Electroencephalogram recordings | 12 weeks
  Power spectra between 1 and 80 Hz (using the Fourier basis with a 2 s wide Hanning window) will be calculated based on clean data from all sensors (electrodes).
Electroencephalogram recordings | 12 weeks
  The average power of each classical frequency band (delta (1-4 Hz), theta (4.1-8 Hz), alpha (8.1-12 Hz), beta (12.1-32 Hz), and gamma (32.1-80 Hz). These measures will be used to test for differences in basic EEG parameters across conditions (rest, Montreal Imaging Stress Task (MIST)) and groups (early, middle and late timepoints), as well as for correlations with key demographic and clinical variables.
Electroencephalogram recordings | 12 weeks
  Time Frequency Analysis: For EEG data acquired during the Montreal Imaging Stress Task (MIST), we will also quantify continuous changes in power of EEG frequency bands as a function of time (i.e., prior to, during and after the Montreal Imaging Stress Task (MIST)).

OTHER OUTCOMES:
Depression, Anxiety, and Stress Scale - 21 (DASS-21) | 12 weeks
  The DASS 21 is a 21-item self-report questionnaire designed to measure the severity of a range of symptoms common to both Depression and Anxiety. In completing the DASS, the individual is required to indicate the presence of a symptom over the previous week. Each item is scored from 0 (did not apply to me at all over the last week) to 3 (applied to me very much or most of the time over the past week).
  The DASS subscores Depression: ranges from 0-9 (normal) to 28+ (extremely severe depression) Anxiety: Ranges from 0-7 (normal) to 20+ (extremely severe anxiety) Stress: Ranges from 0-14 (normal) to 34+ (extremely severe stress)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Cade, BSc, BSc(chiro), MHSc, PhD, Principal Investigator — Scotland College of Chiropractic
Locations (1):
- Scotland College of Chiropractic, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, anonymised post-process eeg data will be made available
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 01/10/2024 for up to two years (01/10/2026)
Access Criteria: Other researchers Via emailing the chief investigator